CLINICAL TRIAL: NCT03036059
Title: Cluster Randomized Community-based Trial of Annual Versus Biannual Single-dose Ivermectin Plus Albendazole Against Wuchereria Bancrofti Infection in Human and Mosquito Populations
Brief Title: Twice Yearly Treatment for the Control of LF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Noguchi Memorial Institute for Medical Research (Other)
Collaborators: Ghana Health Services (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMA 2015 CDF - 976
Record Dates: First submitted 2016-11-03; First posted 2017-01-30 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2018-03

CONDITIONS: Lymphatic Filariasis; Helminth Infection
Keywords: Twice a year treatment; Biannual treatment; Wuchereria bancrofti
MeSH Terms: conditions — Elephantiasis, Filarial; Trematode Infections | interventions — Ivermectin; Albendazole

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): 400 μg/kg Ivermectin + 400 mg Albendazole Tablets given every year for 2 years
  Interventions: Drug: 400 μg/kg Ivermectin + 400 mg Albendazole
- Expanded frequency group (Experimental): 400 μg/kg Ivermectin + 400 mg Albendazole, Tablets given every 6 months for 2 years
  Interventions: Drug: 400 μg/kg Ivermectin + 400 mg Albendazole

INTERVENTIONS:
Drug: 400 μg/kg Ivermectin + 400 mg Albendazole — 400ug/Kg, tablet, given orally once or twice a year.
  Other Names: Mectizan, Stromectol

SUMMARY:
The Global Program for the Elimination of Lymphatic Filariasis (GPELF) has been in operation sing the year 2000, with the aim of eliminating the disease by the year 2020, following 5-6 rounds of effective annual Mass Drug Administration (MDA). The treatment regimen is Ivermectin (IVM) in combination with Diethylcarbamazine (DEC) or Albendazole (ALB). In Ghana, MDA has been undertaken since 2001. While the disease has been eliminated in many areas, transmission has persisted in some implementation units that had experienced 15 or more rounds of MDA. Alternative intervention strategies, including twice yearly MDA and sleeping under insecticidal nets have significantly accelerated transmission interruption in some settings of high transmission intensity. Thus, it is evident that new intervention strategies could eliminate residual infection in areas of persistent transmission and speed up the LF elimination process. This study therefore seeks to test the hypothesis that biannual treatment of LF endemic communities will accelerate interruption of LF transmission.

Two cluster randomized trials will be implemented in LF endemic communities in Ghana. The interventions will be yearly or twice-yearly MDA delivered to entire endemic communities. Allocation to study group will be by clusters identified using the prevalence of LF. Clusters will be randomised to one of two groups: receiving either (1) annual treatment with IVM+ALB; (2) annual MDA with IVM +ALB, followed by an additional MDA 6 months later. The primary outcome measure is the prevalence of LF infection, assessed by four cross-sectional surveys. Entomological assessments will also be undertaken to evaluate the transmission intensity of the disease in the study clusters. Costs and cost-effectiveness will be evaluated. Among a random subsample of participants, microfilaria prevalence will be assessed longitudinally. A nested process evaluation, using semi-structured interviews, focus group discussions and a stakeholder analysis, will investigate the community acceptability, feasibility and scale-up of each delivery system.

ELIGIBILITY:
Inclusion Criteria:

* Residency in the disease endemic community for at least 12 months
* Willingness to provide informed consent/assent
* Willingness to donate blood (per the protocol)

Exclusion Criteria:

* Recent residents (<12 months)
* Inability to give informed consent
* Pregnant and lactating women
* Children below the age of 5.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1462 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2019-12-08 (Actual); Study Completion 2019-12-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline prevalence of Lymphatic Filariasis at 24 months | 0 and 24 months
  The primary outcome, the prevalence of LF infection, will be measured through cross-sectional parasitological surveys conducted at baseline and at 24 months. The timing of the final follow-up survey will take into account differences in time since treatment of the annual and biannual treatment groups at 24 months

SECONDARY OUTCOMES:
Longitudinal assessment of transmission dynamics of Lymphatic Filariasis for modelling the impact of treatment | 0, 12, 24, 30 months
  For the secondary outcome, a subsample of individuals from the clusters in each of the study groups will be followed longitudinally for two and half years, in order to better understand the transmission dynamics of LF and to estimate key parameters for mathematical modelling of transmission dynamics and treatment impact.
Evaluation of community acceptability of twice-yearly treatment, through questionnaires and focus group discussions | 24 months
  A process evaluation, using semi-structured interviews, focus group discussions (FGDs) and a stakeholder analysis, will investigate the community acceptability of the twice-yearly drug administration.
Feasibility of scale-up of twice-yearly treatment, through questionnaires and focus group discussions | 24 months
  A process evaluation, using semi-structured interviews, focus group discussions (FGDs) and a stakeholder analysis, will investigate the feasibility of scaling up the twice-yearly drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Dziedzom K de Souza, PhD, Principal Investigator — Noguchi Memorial Institute for Medical Research
Locations (1):
- Noguchi Memorial Institute for Medical Research, Legon-Accra, Ghana

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared publicly. Researchers interested in the data can contact the principal investigator directly. No personal identifying information will be shared.

REFERENCES:
- [Derived] de Souza DK, Ahorlu CS, Adu-Amankwah S, Otchere J, Mensah SK, Larbi IA, Mensah GE, Biritwum NK, Boakye DA. Community-based trial of annual versus biannual single-dose ivermectin plus albendazole against Wuchereria bancrofti infection in human and mosquito populations: study protocol for a cluster randomised controlled trial. Trials. 2017 Oct 2;18(1):448. doi: 10.1186/s13063-017-2196-9. PMID 28969715